CLINICAL TRIAL: NCT03326336
Title: A Phase 1/2a, Open-Label, Non-Randomized, Dose-Escalation Study to Evaluate the Safety and Tolerability of GS030 in Subjects With Retinitis Pigmentosa
Brief Title: Dose-escalation Study to Evaluate the Safety and Tolerability of GS030 in Subjects With Retinitis Pigmentosa
Acronym: PIONEER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS030_CLIN_001; 2017-002204-27 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2017-10-31 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Non-syndromic Retinitis Pigmentosa
Keywords: Eye Diseases; Hereditary Eye Diseases; Retinal degeneration; Inherited retinal diseases; Rod & cone dystrophies; Retinitis Pigmentosa; Gene Therapy; Optogenetic; Intravitreal Injections; AAV Vectors; Medical device; Visual Interface
MeSH Terms: conditions — Eye Diseases; Eye Diseases, Hereditary; Retinal Degeneration; Cone-Rod Dystrophies; Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: 3 dose-escalation cohorts with 3 subjects per each cohort plus 1 extension cohort at the highest well-tolerated dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cohort (Other): 3 dose escalation cohorts (low, medium and high dose) with 3 subjects per cohort followed by an extension cohort at the highest-well tolerated dose with 3 to 9 subjects.
  Interventions: Combination Product: Gene therapy: GS030-DP AND Medical device: GS030-MD

INTERVENTIONS:
Combination Product: Gene therapy: GS030-DP AND Medical device: GS030-MD — GS030-Drug Product (GS030-DP) - Recombinant adeno-associated viral vector, derived from serotype 2 (rAAV2.7m8), containing the optimized channelrhodopsin ChrimsonR-tdTomato gene under the control of the ubiquitous CAG promoter (rAAV2.7m8-CAG-ChrimsonR-tdTomato) GS030-Medical Device (GS030-MD) - Visual Interface Stimulating Glasses (that amplify the external visual stimulus to the optogenetically engineered retina)

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of escalating doses of a gene therapy called GS030-DP (injected study treatment) administered via a single intravitreal injection and repeated light stimulation using a medical device called GS030-MD (stimulating glasses) in subjects with documented diagnosis of non-syndromic Retinitis Pigmentosa

DETAILED DESCRIPTION:
Study GS030_CLIN_001 is a multicenter, Phase 1/2a, open-label, non-randomized, dose-escalation, safety and tolerability study of GS030-DP in association with GS030-MD in subjects with non-syndromic RP that is confirmed by full-field ERG. The study design includes a dose escalation of the vector encoding the ChR-tdT. This first-in-human study design evaluates the safety and tolerability of GS030, the associated GS030-MD and GS030-DP, which is the treatment to be developed and considered for marketing.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years to ≤75 years at the time of ICF signature.
* Diagnosis of non-syndromic RP defined as:

  * Clinical diagnosis of non-syndromic RP based on history, mid-peripheral visual dysfunction, and fundoscopic appearance.
  * Diagnosis of non-syndromic RP is confirmed on full-field ERG
* Visual acuity:

  * Visual acuity in the dose-escalation cohorts of no better LP.
  * Visual acuity in the extension cohort of no better than CF pending review of dose-escalation cohort data by the DSMB.
* Relatively preserved ganglion cell layer volume and retinal nerve fiber layer thickness, as measured with spectral domain optical coherence tomography (SD-OCT).
* Interpupillary distance of ≥51 mm and ≤72 mm.
* Refractive error of the study eye between -6 diopters and +6 diopters.

Exclusion criteria

* Prior receipt of any gene therapy.
* Subjects who have undergone significant ocular surgery (per investigator determination) within 3 months prior to Visit 1.
* Presence of narrow iridocorneal angles contraindicating pupillary dilation.
* Presence of disorders of the ocular media which interfere with visual acuity and other ocular assessments, including SD-OCT, during the study period.
* Presence of any systemic or ocular diseases, or pathologies, other than non-syndromic RP, or their associated therapies, that can cause or have the potential to cause vision loss.
* Prior vitrectomy or vitreomacular surgery.
* Presence of vitreo-macular adhesion or traction, epiretinal membrane, macular pucker and macular hole, evident by ophthalmoscopy and/or by SD-OCT examinations and assessed by the investigator to significantly affect central vision.
* Current evidence of retinal detachment assessed by the investigator to significantly affect central vision.
* Active ocular inflammation or recurrent history of idiopathic or autoimmune associated uveitis.
* Presence of an Active Implantable Medical Device.
* Subjects who have undergone thermal laser procedure to the retina within 3 months of trial entry, or any prior thermal laser procedure to the macular region.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-10-26 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of escalating doses of GS030-DP administered via a single IVT and repeated light stimulation using GS030-MD in subjects with non-syndromic Retinitis Pigmentosa | Week 52/Year 1
  Safety and tolerability of GS030 treatment at Week 52/Year 1, by assessments based on local and systemic safety issues, specifically those related to IVT of GS030-DP and the subsequent repeated use of GS030-MD, as assessed by incidence of Adverse Events.

SECONDARY OUTCOMES:
Evaluate the treatment effect of GS030 as assessed by visual acuity | Week 52/Year 1
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with the Freiburg Visual Acuity & Contrast Test (FrACT) free computer program that uses graphics capabilities and psychometric methods to provide automated, self-paced measurement and the full field threshold stimulus test (FST) measuring the illuminance necessary to stimulate the most sensitive parts of the retina, and thus determines a quantifiable stimulation threshold (before and after gene transfer, with GS030-MD turned ON and turned OFF).
Evaluate the treatment effect of GS030 as assessed by visual function | Week 52/Year 1
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Humphrey visual field 10-2 Standardized automated perimetry, square localization test, displaying white square at a random location on a black background and direction of motion test measuring the ability of subjects to determine the direction of an object moving in the visual field (before and after gene transfer, with GS030-MD turned ON and turned OFF).
Evaluate the treatment effect of GS030 as assessed by mobility (door task). | Week 52/Year 1
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with door task (before and after gene transfer, with GS030-MD turned ON and turned OFF).
Evaluate the treatment effect of GS030 as assessed by mobility (line task). | Week 52/Year 1
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with line task (before and after gene transfer, with GS030-MD turned ON and turned OFF).
Evaluate the treatment effect of GS030 as assessed by QoL (VFQ25) | Week 52/Year 1
  Assessment of the treatment effect on quality of life changes from baseline to Week 52 with the Visual Functioning Questionnaire-25 (VFQ-25). VFQ25 is a 25-item questionnaire with 47 questions, each question has several responses scored on a scale from 0 to 5, 0 to 6, or 0 to 10. Values are calculated in percentages.
Evaluate the treatment effect of GS030 as assessed by QoL (SF36) | Week 52/Year 1
  Assessment of the treatment effect on quality of life changes from baseline to Week 52 with the Short Form Survey 36 Version 2 (SF-36v2). The SF-36v2 is a subject-rated 36-item questionnaire assessing subject health. There are 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0 to 100 scale. A lower score indicates more disability, and a higher score indicates less disability (a score of 0 is equivalent to maximum disability, and a score of 100 is equivalent to no disability).
Evaluate immune response to recombinant adeno associated viral vector, derived from serotype 2 (rAAV2.7m8) and ChR tdT protein. | Week 52/Year 1
  Immune response to rAAV2.7m8 and ChR-tdT protein from baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Magali Taiel, MD, Study Director — GenSight Biologics
Locations (3):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States
- Centre Hospitalier National d'Ophtalmologie (CHNP) des Quinze-Vingts, Paris, France
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

REFERENCES:
- See also: Website of GenSight Biologics — http://www.gensight-biologics.com/